CLINICAL TRIAL: NCT00122226
Title: MEDICLAS Study (Metabolic Effects of Different Classes of AntiretroviralS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Abbott (Industry); Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: protocol 02-72
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2006-04-25 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections; HIV-Associated Lipodystrophy Syndrome
Keywords: HIV; HIV-associated lipodystrophy syndrome
MeSH Terms: conditions — HIV Infections; HIV-Associated Lipodystrophy Syndrome | interventions — Lopinavir; Ritonavir; Zidovudine; Lamivudine; Nevirapine

INTERVENTIONS:
Drug: Lopinavir/ritonavir + zidovudine + lamivudine
Drug: Lopinavir/ritonavir + nevirapine

SUMMARY:
This is a randomized prospective study into metabolic adverse events during different types of initial antiretroviral therapy in HIV-1-infected men.

DETAILED DESCRIPTION:
This is a randomized prospective study into metabolic adverse events during initial antiretroviral therapy in HIV-1-infected men. The following regimens are compared: lopinavir-ritonavir + Combivir and lopinavir-ritonavir + nevirapine (nucleoside reverse transcriptase inhibitor [NRTI]-sparing). Prior to the start of therapy and 3, 12, 24, and 36 months thereafter the distribution of body fat and bone density (bioelectrical impedance analysis [BIA], computed tomography [CT] and dual energy x-ray absorptiometry [DEXA]), lipid spectrum, mitochondrial DNA (peripheral blood mononuclear cells [PBMCs] and adipose tissue biopsies) and vascular measurements are performed. In addition, insulin sensitivity is measured in a subgroup of sixteen individuals by using a hyperinsulinemic euglycemic clamp and performing microvascular measurements. The aim of the study is to obtain prospective insight into the occurrence of various aspects of metabolic adverse events on the one hand and to compare an NRTI-containing therapy with an NRTI-sparing therapy on the other hand. The hypothesis is that in the NRTI-sparing arm, less metabolic and vascular changes are observed than in the NRTI containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 70 years.
* No prior use of antiretroviral therapy
* Indication for antiretroviral treatment according to common standards

Exclusion Criteria:

* Female sex
* Body mass index (kg/m2) > 35.
* Known history of diabetes mellitus or hyperlipidemia
* Use of coenzyme A reductase inhibitor or fibric acid derivative in the last 6 weeks before inclusion
* Use of the following medication: systemic corticosteroids, thiazide diuretics, calcium-entry blockers, angiotensin-converting inhibitors, nitrates
* Use of nandrolone or testosterone
* Any disorder or condition which can be expected to lead to lessened compliance with the study protocol.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2008-07

PRIMARY OUTCOMES:
insulin resistance (3, 12, 24, 36 months)
microvascular function (3, 12, 24, 36 months)
lipid profile (3, 12, 24, 36 months)
body composition (3, 12, 24, 36 months)
macrovascular function (12, 24, 36 months)

SECONDARY OUTCOMES:
mitochondrial DNA in PBMC and fatty tissue (12, 24, 36 months)
gene expression, markers of mitochondrial toxicity, inflammation, apoptosis, fat cell differentiation in fatty tissue (12, 24, 36 months)
bone mineral density (12, 24, 36 months)
natural killer cells (3, 12, 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: S. A. Danner, MD, PhD, Principal Investigator — Free University Medical Center; P. Reiss, MD, PhD, Principal Investigator — Academic Medical Center, National AIDS Therapy Evaluation Centre
Locations (13):
- Helsinki University Central Hospital, Helsinki, Finland
- Netherlands (10):
  - Academic Medical Center, Amsterdam
  - Medisch Centrum Jan van Goyen, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, location Oosterpark, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, location Prinsengracht, Amsterdam
  - Slotervaart ziekenhuis, Amsterdam
  - VUMC Free University Medical Center, Amsterdam
  - Kennemer Gasthuis, location Elisabeth, Haarlem
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Universitair Medisch Centrum, Rotterdam
  - Ziekenhuis Leyenburg, The Hague
- Hospital Clinic, Barcelona, Spain
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] van Vonderen MG, Blumer RM, Hassink EA, Sutinen J, Ackermans MT, van Agtmael MA, Yki-Jarvinen H, Danner SA, Serlie MJ, Sauerwein HP, Reiss P. Insulin sensitivity in multiple pathways is differently affected during zidovudine/lamivudine-containing compared with NRTI-sparing combination antiretroviral therapy. J Acquir Immune Defic Syndr. 2010 Feb;53(2):186-93. doi: 10.1097/QAI.0b013e3181c190f4. PMID 19898246
- [Derived] van Vonderen MG, van Agtmael MA, Hassink EA, Milinkovic A, Brinkman K, Geerlings SE, Ristola M, van Eeden A, Danner SA, Reiss P; MEDICLAS study group. Zidovudine/lamivudine for HIV-1 infection contributes to limb fat loss. PLoS One. 2009 May 21;4(5):e5647. doi: 10.1371/journal.pone.0005647. PMID 19479079
- [Derived] van Vonderen MG, Lips P, van Agtmael MA, Hassink EA, Brinkman K, Geerlings SE, Sutinen J, Ristola M, Danner SA, Reiss P. First line zidovudine/lamivudine/lopinavir/ritonavir leads to greater bone loss compared to nevirapine/lopinavir/ritonavir. AIDS. 2009 Jul 17;23(11):1367-76. doi: 10.1097/QAD.0b013e32832c4947. PMID 19424051
- [Derived] van Vonderen MG, Hassink EA, van Agtmael MA, Stehouwer CD, Danner SA, Reiss P, Smulders Y. Increase in carotid artery intima-media thickness and arterial stiffness but improvement in several markers of endothelial function after initiation of antiretroviral therapy. J Infect Dis. 2009 Apr 15;199(8):1186-94. doi: 10.1086/597475. PMID 19275490